CLINICAL TRIAL: NCT05647668
Title: A Prospective Randomized Trial on Laparoscopic Total vs Partial Fundoplication in Patients With Atypical Symptoms of Gastroesophageal Reflux Disease
Brief Title: Laparoscopic Total vs Partial Fundoplication in Patients With Atypical Symptoms of Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mykola Paranyak (Other)
Responsible Party: Sponsor-Investigator, Mykola Paranyak, MD, PhD, assistant professor at the Department of General Surgery, Danylo Halytsky Lviv National Medical University
Organization: Danylo Halytsky Lviv National Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2708A
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic Nissen fundoplication (Active Comparator): Creation of a 360° fundoplication wrap over a 30-Fr intra-esophageal bougie.
  Interventions: Procedure: Laparoscopic fundoplication
- laparoscopic Toupet fundoplication (Active Comparator): Creation of a 270° fundoplication wrap over a 30-Fr intra-esophageal bougie.
  Interventions: Procedure: Laparoscopic fundoplication

INTERVENTIONS:
Procedure: Laparoscopic fundoplication — Creation of either a 360° (in Nissen group) or a 270° (in Toupet group) fundoplication wrap over a 30-Fr intra-esophageal bougie.

SUMMARY:
One hundred and twenty patients with documented extraesophageal symptoms of gastroesophageal reflux disease were randomized to either undergo floppy Nissen (n= 60) or Toupet fundoplication (n= 60). Symptom scores of extraesophageal symotoms and quality of life were prospectively evaluated. Analysis of the treatment results showed a significant improvement of symptoms in both patient groups.Quality of life improved substantially at short- and long-term follow up in both groups and there were no statistical differences between the groups in this parameter.

ELIGIBILITY:
Inclusion Criteria:

* extraesophageal symptoms of gastroesophageal reflux disease
* undergoing surgery for gastroesophageal reflux disease
* at least 18 years old

Exclusion Criteria:

* patients under the age of 18 years
* previous anti-reflux surgery, other surgical procedures in the vicinity of the gastroesophageal junction
* major psychiatric illness
* unstable chronic illnesses (such as diabetes)
* inability of the patient to complete the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Symptom scores of throat clearing, globus sensation, cough, throat pain, vocal changes. | 24 month

SECONDARY OUTCOMES:
Reflux symptom index (RSI) score | 24 months
  The reflux symptom index (RSI) questionnaire is a nine-item, 45-point survey used in the evaluation of symptoms of laryngopharyngeal reflux. A RSI score higher than 13 is considered abnormal and indicates the presence of laryngopharyngeal reflux.
laryngopharyngeal reflux-health-related quality of life (LPR-HRQL) questionnaire score | 24 months
  The LPR-HRQL questionnaire is a 43-item survey, designed to assess the effects of extraesophageal reflux symptoms on social and occupational functioning, vitality, well-being and perceived health.

CONTACTS AND LOCATIONS:
Locations (1):
- Danylo Halytsky Lviv National Medical University, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided after publication of the article